CLINICAL TRIAL: NCT06178211
Title: Neoadjuvant Adebrelimab Plus Chemotherapy for Resectable ESCC: a Single Arm, Prospective Phase 2 Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief of Department of Esophageal Surgery, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-015
Record Dates: First submitted 2023-11-18; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adebrelimab and chemotherapy (Experimental)
  Interventions: Drug: Immunotherapy: Adebrelimab; Drug: chemotherapy: carboplatin plus nab-paclitaxel

INTERVENTIONS:
Drug: Immunotherapy: Adebrelimab — Adebrelimab 1200mg Q3W
Drug: chemotherapy: carboplatin plus nab-paclitaxel — carboplatin plus nab-paclitaxel

SUMMARY:
The investigators will conduct a single-arm prospective study to evaluate the efficacy and safety of neoadjuvant therapy with adebrelimab (SHR-1316) and chemotherapy in patients with resectable esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects signed the informed consent and volunteered to participate in the study.
2. Esophageal squamous cell carcinoma confirmed by histology or cytology.
3. Thoracic esophageal squamous cell carcinoma confirmed by CT or pet-CT, which is classified as cII-III (AJCC 8th).
4. Expect to have R0 resection
5. In age from 18 to 75.
6. ECOG PS: 0~1.
7. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, etc.
8. No contraindications to surgery.
9. Has sufficient organ function including (1) Blood routine: NE≥1.5×109/L; PLT≥100×109/L; HGB≥90 g/L (2)Comprehensive Metabolic Panel: bilirubin≤ 1.5×ULN; ALT≤2.5×ULN; AST≤2.5×ULN; sCr≤1.5×ULN or CrCl≥50 mL/min（Cocheroft-Gault) (3) Coagulation function: INR≤1.5; APTT≤1.5×ULN
10. Women of childbearing age must undergo a serological pregnancy test within 72 hrs before first administration. Women of childbearing age, or male subjects with childbearing age female partners, must take contraceptive measures from the first dose to three months after last administration.
11. Good compliance, willing to comply with follow-up schedules.

Exclusion Criteria:

1. Subjects have received or are receiving any of:

   1. anti-tumor interventions such as radiotherapy, chemotherapy or other medictions.
   2. immunosuppresants or systemic glucosteroids (prednisone equivalence> 10mg/d) within 2 weeks before the first administration, inhaled or topical use of glucosteroids (prednisone equivalence>10mg/d) is allowed if no known active autoimmune disease.
   3. live vaccine within 4 weeks before the first administration.
   4. major surgery or major injury within 4 weeks before the first administration.
2. Cancer related exclusion criteria

   1. other cancers instead of ESCC
   2. non-recetable or metastatic ESCC
   3. not comply with cⅡ-Ⅲ（cT2N1-2M0 or cT3N0-2M0, AJCC 8th）
   4. Subjects with other malignant tumors within 5 years before the first administration, but subjects with cervical carcinoma in situ, skin basal cell carcinoma, skin squamous cell carcinoma, localized prostate cancer received radical surgery and ductal carcinoma in situ that have received radical treatment and do not need other treatment can be included)
3. Other criteria

   1. Subjects have uncontrolled cardiovascular diseases, such as 1) heart failure ≥ NYHA class 2, 2) unstable angina 3) myocardial infarction within 1 year; 4) supraventricular or ventricular arrthymia that needs treatment
   2. Subjects with any known active autoimmune disease
   3. Pregnant or breastfeeding female
   4. Presence of allergy or hypersensitivity to investigational medications
   5. HIV positive or active hepatitis B (HbsAg positive and HBV-DNA ≥2000 IU/ml or ≥ 104 copies/mL) or active hepatitis C (HCV antibody positive) or active tuberculosis
   6. Investigators assessed there might be other factors that cause subjects to withdrawl.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 12 months
  The primary endpoint is a pCR rate, which is defined as the absence of any remaining tumor cells in both the main tumor and the nearby lymph nodes (ypT0N0) as per the AJCC 8th Edition TRG scoring system.

SECONDARY OUTCOMES:
cCR rate | 12 months
  A clinical complete response rate (cCR) is defined as the complete disappearance of tumor lesions as assessed by enhanced CT, endoscopic ultrasound, and endoscopic biopsy.
R0 resection rate | 12 months
  A R0 resection rate is defined as the rate of complete tumor removal with negative resection margin microscopically
MPR rate | 12 months
  A major pathological response rate (MPR) is defined as the proportion of residual living tumor cells in the post-surgery specimen within the tumor bed being less than or equal to 10%.
median EFS | 12 months
  An event-free survival (EFS) is defined as the duration from the start of treatment until disease recurrence or death from any cause, whichever occurs first.
median OS | 12 months
  An overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence.
Incidence, type and severity of adverse events as assessed by CTCAE 5.0 | From date of treatment allocation until surgery was applied during study period or up to at least 90 days after last dose
  Including adverse events and complications. Incidence of adverse events using CTCAE 5.0; grade 3 treatment-related adverse events and higher-grade will be reported
Potential biomarkers such as ctDNA or PD-L1 expression | 12 months
  Potential biomarkers such as ctDNA or PD-L1 expression will be explored and analysed using blood or tissues prior and post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided